CLINICAL TRIAL: NCT01302119
Title: A Randomized, Double-Blind, Vehicle-Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of AN2690 Topical Solution, 5%, vs. Solution Vehicle in the Treatment of Onychomycosis of the Toenail in Adults
Brief Title: Efficacy and Safety of AN2690 Topical Solution to Treat Onychomycosis of the Toenail
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN2690-ONYC-302
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Onychomycosis of Toenails
Keywords: Onychomycosis; nail fungus; toenail fungus; fungal nail; hyperkeratosis; nail infection; nail treatment; toenail infection; toenail treatment; foot dermatoses; fungal culture; onycholysis; podiatrist; podiatry; subungual; tinea unguium; antifungal; anti-fungal; dermatologist; dermatology; dermatophyte; distal subungual onychomycosis; yellow nail; thick nail; brittle nail; crumbling nail; discolored nail; weak nail
MeSH Terms: conditions — Onychomycosis; Keratoderma, Palmoplantar, Epidermolytic; Foot Dermatoses; Onycholysis; Yellow Nail Syndrome; Nails, Malformed; Twenty-Nail Dystrophy | interventions — Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AN2690 Topical Solution, 5% (Experimental): AN2690 Topical Solution, 5%
  Interventions: Drug: AN2690 Topical Solution, 5%
- Solution Vehicle (Placebo Comparator): Solution Vehicle
  Interventions: Drug: Solution Vehicle

INTERVENTIONS:
Drug: AN2690 Topical Solution, 5% — AN2690 Topical Solution, 5%, applied once daily for 48 weeks
  Arms: AN2690 Topical Solution, 5%
Drug: Solution Vehicle — AN2690 Topical Solution, Vehicle, applied once daily for 48 weeks
  Arms: Solution Vehicle

SUMMARY:
The purpose of this study is to determine whether AN2690 topical solution is a safe and effective treatment for onychomycosis of the toenail.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of distal subungual onychomycosis affecting at least one great toenail
* KOH positive at screening
* Willingness not to use any other products including nail polish applied to the toenails during the study
* Women of childbearing potential who are currently sexually active must agree to use contraception for the entire study period

Exclusion Criteria:

* Concurrent or recent use of certain topical or systemic medications without a sufficient washout period
* History of any significant chronic fungal disease other than onychomycosis
* Significant confounding conditions as assessed by study doctor
* Participated in any other trial of an investigational drug or device within 30 days or participation in a research study concurrent with this study
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12-31 (Actual); Study Completion 2013-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PfizerCT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (25):
  - Investigational Site, Phoenix, Arizona
  - Investigational Site, Novato, California
  - Investigational Site, Oceanside, California
  - Investigational Site, San Diego, California
  - Investigational Site, San Francisco, California
  - Investigational Site, Santa Rosa, California
  - Investigational Site, Miami, Florida
  - Investigational Site, Nampa, Idaho
  - Investigational Site, Evansville, Indiana
  - Investigational Site, Ann Arbor, Michigan
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Verona, New Jersey
  - Investigational Site, Albuquerque, New Mexico
  - Investigational Site, High Point, North Carolina
  - Investigational Site, Raleigh, North Carolina
  - Investigational Site, Columbus, Ohio
  - Investigational Site, Portland, Oregon
  - Investigational Site, Philadelphia, Pennsylvania
  - Investigational Site, Greer, South Carolina
  - Investigational Site, Knoxville, Tennessee
  - Investigational Site, Dallas, Texas
  - Investigational Site, San Antonio, Texas
  - Investigational Site, Salt Lake City, Utah
  - Investigational Site, Harrisonburg, Virginia
  - Investigational Site, Norfolk, Virginia
- Canada (6):
  - Investigational Site, Barrie, Ontario
  - Investigational Site, Markham, Ontario
  - Investigational Site, North Bay, Ontario
  - Investigational Site, Boucherville, Quebec
  - Investigational Site, Montreal, Quebec
  - Investigational Site, Québec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at forty-two investigative centers in the United States and Canada. The study population included men and women, 18 years of age and older who had distal subungual onychomycosis. The first subject visit occurred on February 2, 2011, and the last subject completed the Post Study Follow Up on February 20, 2013.
Pre-assignment Details: Eligible subjects were randomized in a 2:1 ratio to receive AN2690 Topical Solution, 5% or Solution Vehicle to be applied once daily to all affected toenails throughout the 48-week treatment period.
Period: Overall Study
Arm/Group | AN2690 Topical Solution, 5% | Solution Vehicle
Started | 399 | 205
Completed | 349 | 177
Not Completed | 50 | 28
Not completed — Withdrawal by Subject | 30 | 20
Not completed — Lost to Follow-up | 10 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Non-compliance | 4 | 2
Not completed — Non-specific | 4 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed using the intent-to-treat (ITT) population. Demographic characteristics were also analyzed using the Per Protocol (PP), Safety, and Post Study Follow Up (PSFU) populations, and were consistent with those of the ITT population. Safety analysis was performed using the Safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | AN2690 Topical Solution, 5% | Solution Vehicle | Total
Number analyzed (Participants) | 396 | 205 | 601
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (11.5) | 55.4 (11.0) | 55.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 31 | 104
  Male | 323 | 174 | 497
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 30 | 87
  Not Hispanic or Latino | 339 | 175 | 514
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 11 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 21 | 14 | 35
  White | 355 | 183 | 538
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 315 | 165 | 480
  Canada | 81 | 40 | 121

OUTCOME MEASURES:

1. Primary Outcome: Complete Cure (Completely Clear Nail and Negative Mycology) of Target Great Toenail at Week 52
Description: No clinical evidence of onychomycosis as evidenced by normal toenail plate, no onycholysis, and no subungual hyperkeratosis, and negative KOH wet mount and negative fungal culture.
Time Frame: Week 52
Population: Efficacy analysis was performed using the ITT population. The last observation was carried forward (LOCF) in order to provide a value for efficacy parameters that were missing.
Measure: Number; unit: participants
Arm/Group | AN2690 Topical Solution, 5% | Solution Vehicle
Number analyzed (Participants) | 396 | 205
participants
  Success | 36 | 3
  Failure | 360 | 202
Statistical Analysis 1: Comparison: AN2690 Topical Solution, 5% vs Solution Vehicle; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Completely Clear or Almost Clear Target Great Toenail at Week 52
Description: No clinical evidence of onychomycosis as evidenced by normal toenail plate, no onycholysis, and no subungual hyperkeratosis, or no more than minimal evidence of onychomycosis as evidenced by toenail plate dystrophic or discolored over ≤ 10% of the distal aspect, with minimally evident onycholysis and subungual hyperkeratosis.
Time Frame: Week 52
Population: Efficacy analysis was performed using the ITT population. The LOCF was used in order to provide a value for efficacy parameters that were missing.
Measure: Number; unit: participants
Arm/Group | AN2690 Topical Solution, 5% | Solution Vehicle
Number analyzed (Participants) | 396 | 205
participants
  Success | 109 | 30
  Failure | 287 | 175
Statistical Analysis 1: Comparison: AN2690 Topical Solution, 5% vs Solution Vehicle; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Treatment Success (Completely Clear or Almost Clear Nail and Negative Mycology) of Target Great Toenail at Week 52
Description: No clinical evidence of onychomycosis as evidenced by normal toenail plate, no onycholysis, and no subungual hyperkeratosis, or no more than minimal evidence of onychomycosis as evidenced by toenail plate dystrophic or discolored over ≤ 10% of the distal aspect, with minimally evident onycholysis and subungual hyperkeratosis, and negative KOH wet mount and negative fungal culture.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | AN2690 Topical Solution, 5% | Solution Vehicle
Number analyzed (Participants) | 396 | 205
participants
  Success | 71 | 8
  Failure | 325 | 197
Statistical Analysis 1: Comparison: AN2690 Topical Solution, 5% vs Solution Vehicle; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Negative Mycology of Target Great Toenail at Week 52
Description: Negative KOH and negative fungal culture.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | AN2690 Topical Solution, 5% | Solution Vehicle
Number analyzed (Participants) | 396 | 205
participants
  Success | 142 | 25
  Failure | 254 | 180
Statistical Analysis 1: Comparison: AN2690 Topical Solution, 5% vs Solution Vehicle; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: An AE was any unfavorable and unintended sign,symptom,or disease temporally associated with the use of the investigational product. A serious AE resulted in death,was life-threatening,required or prolonged in-patient hospitalization,persistent or significant disability/incapacity,resulted in a congenital anomaly,or was an important medical event.
Arm/Group | AN2690 Topical Solution, 5% | Solution Vehicle
Serious Adverse Events (participants affected / at risk) | 7/395 | 2/202
Other Adverse Events (participants affected / at risk) | 88/395 | 48/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AN2690 Topical Solution, 5% (N=395) | Solution Vehicle (N=202)
Retinal artery occlusion (unrelated) (Eye disorders) | 1 | 0
Appendicitis (unrelated) (Infections and infestations) | 1 | 0
Bronchitis (unrelated) (Infections and infestations) | 0 | 1
Cystitis (unrelated) (Infections and infestations) | 1 | 0
Femur fracture (unrelated) (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (unrelated) (Musculoskeletal and connective tissue disorders) | 1 | 0
Carotid artery disease (unrelated) (Nervous system disorders) | 0 | 1
Cerebrovascular accident (unrelated) (Nervous system disorders) | 1 | 0
Transient ischaemic attack (unrelated) (Nervous system disorders) | 0 | 1
Anxiety (unrelated) (Psychiatric disorders) | 1 | 0
Pulmonary embolism (unrelated) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic aneurysm (unrelated) (Vascular disorders) | 0 | 1
Deep vein thrombosis (unrelated) (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (unrelated) (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AN2690 Topical Solution, 5% (N=395) | Solution Vehicle (N=202)
Tinea pedis (Infections and infestations) | 53 | 25
Nasopharyngitis (Infections and infestations) | 27 | 16
Upper respiratory tract infection (Infections and infestations) | 18 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution or Principal Investigator may only publish Study results after: (i) the results of the multicenter Study in its entirety have been publicly disclosed by the Sponsor in an abstract, manuscript or presentation form, or (ii) two (2) years after conclusion of the Study at all sites, whichever is first to occur.